CLINICAL TRIAL: NCT04589741
Title: An Open, Multicenter, Randomized, Phase II Study of Toripalimab Combined With CAV/IE Regimen in Patients With Advanced or Unresectable Bone and Soft Tissue Sarcomas Who Failed Standard Treatment
Brief Title: Toripalimab Combined With CAV/IE Regimen
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xing Zhang, Director of department of medical sarcoma and melanoma,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Toripalimab plus chemotherapy
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- toripalimab combined with CAV/IE regimen (Experimental): toripalimab combined with CAV/IE regimen in patients with advanced or unresectable bone and soft tissue sarcomas who failed standard treatment
  Interventions: Drug: Toripalimab Combined With CAV/IE chemotherapy; Drug: CAV/IE alternate chemotherapy
- CAV/IE chemotherapy alone (Placebo Comparator): CAV/IE chemotherapy alone in patients with advanced or unresectable bone and soft tissue sarcomas who failed standard treatment
  Interventions: Drug: Toripalimab Combined With CAV/IE chemotherapy; Drug: CAV/IE alternate chemotherapy

INTERVENTIONS:
Drug: Toripalimab Combined With CAV/IE chemotherapy — CAV/IE regimen alternate chemotherapy (regimen 1: CTX 1.2mg/m2 D1 + ADM 50mg/m2 D1 + VCR 1.4mg/m2 D1 and scheme 2: IFO 1.5g/m2 D1-5 + vp-16 90mg / m2 D1-5, IV drip). Regimen 1 and 2 were performed alternately, with a cycle of 3 weeks;
  The patients were treated with toripalimab (240mg, 6ml) intravenously every 3 weeks;
  If doxorubicin has reached the upper limit or reduced cardiac toxicity, liposome adriamycin (50mg/m2) or IE regimen can be used
  After 6 courses of treatment, patients with disease control (CR + PR + SD) and tolerable adverse reactions were treated continuously. The study was completed when the researchers considered that the patients were not suitable for continuous medication or the efficacy evaluation was disease progression (PD). No other anti-tumor treatment can be carried out during the treatment.
Drug: CAV/IE alternate chemotherapy — CAV/IE alternate chemotherapy (regimen1: CTX 1.2mg/m2 D1 + ADM 50mg/m2 D1 + VCR 1.4mg/m2 D1 and regimen2: IFO 1.5g/m2 D1-5 + VP-16 90mg/m2 D1-5, IV drip), regimen 1 and 2 were performed alternately, with a cycle of 3 weeks.
  Patiens with disease control (CR+PR+SD) and tolerable adverse reactions were treated continuously with a maximum of 8-10 cycles. If doxorubicin has reached the upper limit or reduced cardiac toxicity, liposome adriamycin (≥ 60 years old: 35mg/m2, < 60 year old: 40mg/m2) or IE regimen can be used. The study was completed when the researchers considered that the patients were not suitable for continuous medication or the efficacy evaluation was disease progression (PD). No other anti-tumor treatment can be carried out during the treatment.

SUMMARY:
The aim of this study was to investigate the efficacy and safety of CAV/IE chemotherapy combined with toripalimab versus CAV/IE chemotherapy alone in the treatment of patients with advanced or unresectable bone and soft tissue sarcomas who failed in standard treatment.

DETAILED DESCRIPTION:
At present, there are many clinical trials of chemotherapy drugs combined with anti-PD-1 antibody in the treatment of tumor, but the clinical study of CAV/IE chemotherapy combined with anti-PD-1 antibody in the treatment of advanced or non resectable bone and soft tissue sarcoma has not been started, and the related research is still in the blank state. In view of the above problems, to observe and evaluate the efficacy and safety of CAV/IE chemotherapy combined with toripalimab versus CAV/IE chemotherapy alone in the treatment of advanced or non resectable bone and soft tissue sarcoma patients, so as to provide more treatment options for patients with advanced or non resectable bone and soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study and signed informed consent;

   For all advanced or non resectable bone and soft tissue sarcomas confirmed by pathology, the standard treatment failed or there was no standard treatment. They were mainly synovial sarcoma, leiomyosarcoma, undifferentiated pleomorphic sarcoma, liposarcoma, fibrosarcoma, clear cell sarcoma, angiosarcoma, epithelioid sarcoma, malignant peripheral nerve sheath tumor, undiffertiated sarcoma, bone sarcoma, chondrosarcoma, Ewing's sarcoma, rhabdomyosarcoma, dermatofibrosarcoma protuberans, myofibroblastic sarcoma, malignant solitary fibroma, postradiation sarcoma,etc. But the pathological subtypes without standard treatment can be treated as first-line treatment, including but not limited to postradiation sarcoma, dedifferentiated / pleomorphic liposarcoma, clear cell sarcoma, etc., except for the following types: well differentiated liposarcoma, malignant mesothelioma, gastrointestinal stromal tumor, etc;
2. Advanced patients with unresectable lesions or lymph nodes or distant metastasis assessed by imaging;
3. In the past three months, there was at least one measurable target lesion according to RECIST version 1.1 standard, and it can be accurately measured by magnetic resonance imaging (MRI) or computer tomography (CT) in at least one direction (the maximum diameter needs to be recorded), with conventional CT ≥ 20 mm or spiral CT ≥ 10 mm.
4. They were 14-70 years old; ECOG PS score: 0-1; the expected survival time was more than 3 months;
5. Within 7 days before treatment, the main organ functions met the following criteria:

(1) Blood routine examination standard (without blood transfusion within 14 days)

① Hemoglobin (HB) ≥ 90g / L;

* The absolute value of neutrophil (ANC) ≥ 1.5 × 109 / L;

  * Platelet (PLT) ≥ 80 × 109 / L.

    (2) Biochemical examination should meet the following standards:

    ① Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal value (ULN);
* Alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5uln; ALT and AST ≤ 5uln with liver metastasis

  ③ Serum creatinine (CR) ≤ 1.5uln or creatinine clearance rate (CCR) ≥ 60ml / min;

  (3) Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ the lower limit of normal value (50%).

  6)Women of childbearing age should agree that contraceptive measures (such as intrauterine device, contraceptive or condom) must be used during the study period and within 6 months after the end of the study; serum or urine pregnancy test negative within 7 days before study enrollment, and must be non lactating patients; men should agree that contraceptive measures must be used during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

1) Patients who had previously received anti-PD-1 / PD-L1 antibody therapy.

2) Other malignancies occurred or were present within 5 years, except for cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [ta (non invasive tumor), tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];

3) The patients with thyroid dysfunction after the best drug treatment;

4) Systemic anti-tumor therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or mitomycin C within 6 weeks prior to the trial drug treatment) was planned within 4 weeks before enrollment or during the study period. Over extended field radiotherapy was performed within 4 weeks before admission or limited field radiotherapy was performed within 2 weeks before grouping;

5) With pleural effusion or ascites, it causes respiratory syndrome (≥ CTC AE grade 2 dyspnea [grade 2 dyspnea refers to shortness of breath with a small amount of activity; it affects instrumental activities of daily living]);

6) Any unrelieved toxic reaction higher than CTC AE (4.01) grade 1 or above caused by previous treatment, excluding alopecia;

7) Patients with any severe and / or uncontrolled disease, including:

1. Patients with poor blood pressure control (SBP ≥ 150 mmHg, DBP ≥ 100 mmHg);
2. Patients with myocardial ischemia or myocardial infarction of grade I or above, arrhythmia (including QTc ≥ 480ms) and congestive heart failure (NYHA) grade ≥ 2;
3. Active or uncontrolled severe infection (≥ CTC AE Level 2 infection);
4. Chronic liver disease, decompensated liver disease or decompensated hepatitis;
5. Renal failure needs hemodialysis or peritoneal dialysis;
6. Poor control of diabetes mellitus (FBG > 10mmol / L);
7. Urine routine examination showed that urine protein was ≥ + +, and 24-hour urine protein was more than 1.0 G;
8. Patients with epilepsy and need treatment;

8) Major surgical treatment, open biopsy or obvious traumatic injury were performed within 28 days before admission;

9) Patients with any physical signs or history of bleeding regardless of severity; patients with any bleeding or bleeding events ≥ CTCAE 3 within 4 weeks before enrollment had unhealed wounds, ulcers or fractures;

10) Patients who had AVT events within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;

11) There were active ulcer, intestinal perforation and intestinal obstruction;

12) Subjects with clinical symptoms of central nervous system metastasis (such as brain edema, need for hormone intervention, or brain metastasis progression); patients who have previously received treatment for brain or meningeal metastasis, such as clinical stability (MRI) for at least 2 months, and who have stopped systemic hormone therapy (dose > 10mg / day, prednisone or other effective hormones) for more than 2 weeks can be included;

13) The subjects were using immunosuppressive agents, or systemic or absorbable local hormone therapy to achieve the purpose of immunosuppression (dosage > 10mg / D, prednisone or other effective hormones), and continued to use them within 2 weeks before enrollment;

14) Subjects with any active autoimmune disease or history of autoimmune diseases (e.g., but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; if the subject has vitiligo or asthma has been completely relieved in childhood, it is not necessary to be an adult Any intervention can be included; asthma patients who need bronchodilator for medical intervention cannot be included);

15) The subjects had active tuberculosis;

16) According to the judgment of the researcher, the subjects are not suitable to be enrolled or there are other factors that may lead to termination of the study, such as other serious diseases (including mental diseases) requiring combined treatment, serious laboratory examination abnormalities, and family or social factors, which will affect the safety of the subjects, or the collection of test data and samples;

17) Patients who participated in other clinical trials of anti-tumor drugs within 28 days before enrollment.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate, ORR | up to 24 months
  The percentage of patients with complete remission and partial remission in patients with evaluable curative effect.

SECONDARY OUTCOMES:
Progression-free survival, PFS | Up to 24 months
  PFS was defined as the time from randomization to objective tumor progression or death.
Disease-free surviva, DFS | Up to 24 months
  DFS is defined as the time from randomization to recurrence of tumor or death.
Overall survival, OS | Up to 24 months
  OS is defined as the time from randomization to death.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Zhang, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China